CLINICAL TRIAL: NCT05172063
Title: Persistent SARS-CoV-2 Infection in Children With Cancer and Impaired Immune Responsiveness
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Children's Cancer Hospital Egypt 57357 (Other)
Collaborators: National Research Centre, Egypt (Other); Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: CCHE-Persistent SARS-CoV-2
Record Dates: First submitted 2021-12-26; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Children With Cancer; SARS-CoV-2 Infection
Keywords: Children; Cancer; SARS-CoV-2; Adaptive Immune Response
MeSH Terms: conditions — COVID-19; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Persistent SARS-CoV-2 Infection Group: Pediatric Cancer patients with persistent SARS-CoV-2 infection
- SARS-CoV-2 Clearance Group: Pediatric Cancer patients who tested negative for SARS-CoV-2 within 14 days of diagnosis.

SUMMARY:
The main goal of this study is to characterize the adaptive immune responses to SARS-CoV-2 infection in a cohort of children with cancer and impaired immune responsiveness and prolonged viral shedding of SARS-CoV-2, and to identify SARS-CoV-2 variants that might arise during poorly controlled virus replication

DETAILED DESCRIPTION:
Although the adaptive immune response plays an important role in improving clinical outcomes of patients infected with SARS2, variability in clinical disease and outcome in patients with SARS2 infection has not been explained by the variation in qualitative and quantitative antiviral immune responses. It has been observed that immunocompromised children shed the virus from the upper respiratory tract for prolonged periods of time, even after the resolution of clinical symptoms. Thus deficits in adaptive immune responses might lead to ineffective control of virus replication and prolonged virus shedding. The proposed studies will define the relationship between adaptive immunity and virus replication/shedding, including the contribution of viral variants that could arise during poorly controlled virus replication in children with ineffective immune responses. The specific aims of the proposed study are: (a) To measure (quantify and qualify) the adaptive immune responses (humoral and cell-mediated immune responses) after infection with SARS-CoV-2 in a cohort of hospitalized children with cancer and impaired immune response. (b) To define the long-term kinetics of the antibody response, cell-mediated immune responses following infection with SARS-CoV-2 in a cohort of hospitalized children with cancer and impaired immune response, and to estimate the duration of protective immunity.(c) to statistically assess whether impaired humoral immunity is associated with prolonged viral replication and shedding (persistence) following infection with SARS-CoV-2 in a cohort of children with cancer and impaired immune response, (d) To genetically trace SARS-CoV-2 mutations, and statistically assess the association between persistent SARS-CoV-2 infection and the frequency of viral mutations and the emergence of viral variants in a cohort of children with cancer and impaired immune response, after their infection with SARS-CoV-2 This will be a prospective, observational cohort study design. The study population will include pediatric and adolescent patients undergoing cancer chemotherapy with a confirmed SARS-CoV-2 infection (PCR Positive). Eligible subjects will be followed prospectively for three months from the time they tested positive for SARS-CoV-2 by PCR. SARS-CoV-2 RNA, antibody, and cell-mediated immune responses will be assessed at specified time points and compared between the children with persistent SARS-CoV-2 infection, and those who cleared SARS-CoV-2 virus. Sequence viral variants in the persistent SARS-COV-2 infected group Assess the association between the emergence of viral variants and mutations and strain virulence and clinical outcome

ELIGIBILITY:
Inclusion Criteria:

1. Children (<18) of both genders undergoing cancer chemotherapy
2. Symptomatic SARS-CoV-2 infection, confirmed by (positive PCR test).
3. Patients with hematologic malignancies (ALL, AML, HL & NHL) on active treatment or under follow up < 3 months from end of treatment protocol

Exclusion Criteria:

1. Children (<18 years) of both genders undergoing cancer chemotherapy with (PCR negative) test result for SARS-CoV-2.
2. Children who are PCR positive but are diagnosed with an immune disorder that may confound the study results.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will include pediatric and adolescent patients undergoing cancer chemotherapy with a confirmed SARS-CoV-2 infection (PCR Positive). We will recruit 30 patients undergoing cancer chemotherapy with a confirmed SARS-CoV-2 infection (PCR Positive). Twenty children with persistent SARS-CoV-2 infection, and 10 children with SARS-CoV-2 clearance within 14 days of diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 antibody titers | Three months
Different subsets of immune cells (neutrophils, dendritic cells, B- and T- lymphocytes) | Three months

SECONDARY OUTCOMES:
Sequence viral variants in the persistent SARS-COV-2 infected group | Three months
Assess the association between the emergence of viral variants and mutations and strain virulence and clinical outcome | Three months

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Diaaeldin Hashem, MBBCh, MSc, Principal Investigator — Children's Cancer Hospital Egypt
Locations (1):
- Children's Cancer Hospital Egypt 57357 Cairo, Egypt, Cairo, Egypt

REFERENCES:
- [Result] Sethuraman N, Jeremiah SS, Ryo A. Interpreting Diagnostic Tests for SARS-CoV-2. JAMA. 2020 Jun 9;323(22):2249-2251. doi: 10.1001/jama.2020.8259. No abstract available. PMID 32374370
- [Result] Avanzato VA, Matson MJ, Seifert SN, Pryce R, Williamson BN, Anzick SL, Barbian K, Judson SD, Fischer ER, Martens C, Bowden TA, de Wit E, Riedo FX, Munster VJ. Case Study: Prolonged Infectious SARS-CoV-2 Shedding from an Asymptomatic Immunocompromised Individual with Cancer. Cell. 2020 Dec 23;183(7):1901-1912.e9. doi: 10.1016/j.cell.2020.10.049. Epub 2020 Nov 4. PMID 33248470
- [Result] Baang JH, Smith C, Mirabelli C, Valesano AL, Manthei DM, Bachman MA, Wobus CE, Adams M, Washer L, Martin ET, Lauring AS. Prolonged Severe Acute Respiratory Syndrome Coronavirus 2 Replication in an Immunocompromised Patient. J Infect Dis. 2021 Jan 4;223(1):23-27. doi: 10.1093/infdis/jiaa666. PMID 33089317
- [Result] Choi B, Choudhary MC, Regan J, Sparks JA, Padera RF, Qiu X, Solomon IH, Kuo HH, Boucau J, Bowman K, Adhikari UD, Winkler ML, Mueller AA, Hsu TY, Desjardins M, Baden LR, Chan BT, Walker BD, Lichterfeld M, Brigl M, Kwon DS, Kanjilal S, Richardson ET, Jonsson AH, Alter G, Barczak AK, Hanage WP, Yu XG, Gaiha GD, Seaman MS, Cernadas M, Li JZ. Persistence and Evolution of SARS-CoV-2 in an Immunocompromised Host. N Engl J Med. 2020 Dec 3;383(23):2291-2293. doi: 10.1056/NEJMc2031364. Epub 2020 Nov 11. No abstract available. PMID 33176080
- [Result] Aydillo T, Gonzalez-Reiche AS, Aslam S, van de Guchte A, Khan Z, Obla A, Dutta J, van Bakel H, Aberg J, Garcia-Sastre A, Shah G, Hohl T, Papanicolaou G, Perales MA, Sepkowitz K, Babady NE, Kamboj M. Shedding of Viable SARS-CoV-2 after Immunosuppressive Therapy for Cancer. N Engl J Med. 2020 Dec 24;383(26):2586-2588. doi: 10.1056/NEJMc2031670. Epub 2020 Dec 1. No abstract available. PMID 33259154
- [Result] Truong TT, Ryutov A, Pandey U, Yee R, Goldberg L, Bhojwani D, Aguayo-Hiraldo P, Pinsky BA, Pekosz A, Shen L, Boyd SD, Wirz OF, Roltgen K, Bootwalla M, Maglinte DT, Ostrow D, Ruble D, Han JH, Biegel JA, Li M, Huang C, Sahoo MK, Pannaraj PS, O'Gorman M, Judkins AR, Gai X, Dien Bard J. Increased viral variants in children and young adults with impaired humoral immunity and persistent SARS-CoV-2 infection: A consecutive case series. EBioMedicine. 2021 May;67:103355. doi: 10.1016/j.ebiom.2021.103355. Epub 2021 Apr 26. PMID 33915337
- [Result] Turner JS, Day A, Alsoussi WB, Liu Z, O'Halloran JA, Presti RM, Patterson BK, Whelan SPJ, Ellebedy AH, Mudd PA. SARS-CoV-2 Viral RNA Shedding for More Than 87 Days in an Individual With an Impaired CD8+ T Cell Response. Front Immunol. 2021 Jan 8;11:618402. doi: 10.3389/fimmu.2020.618402. eCollection 2020. PMID 33488630
- [Result] Gomaa MR, Kandeil A, Mostafa A, Roshdy WH, Kayed AE, Shehata M, Kutkat O, Moatasim Y, El Taweel A, Mahmoud SH, Kamel MN, Abo Shama NM, El Sayes M, El-Shesheny R, Bakheet OH, Elgohary MA, Elbadry M, Nassif NN, Ahmed SH, Abdel Messih IY, Kayali G, Ali MA. Prevalence of Severe Acute Respiratory Syndrome Coronavirus 2 Neutralizing Antibodies in Egyptian Convalescent Plasma Donors. Front Microbiol. 2020 Nov 24;11:596851. doi: 10.3389/fmicb.2020.596851. eCollection 2020. PMID 33329484
- [Result] Gomaa MR, El Rifay AS, Shehata M, Kandeil A, Nabil Kamel M, Marouf MA, GabAllah M, El Taweel A, Kayed AE, Kutkat O, Moatasim Y, Mahmoud SH, Abo Shama NM, El Sayes M, Mostafa A, El-Shesheny R, McKenzie PP, Webby RJ, Kayali G, Ali MA. Incidence, household transmission, and neutralizing antibody seroprevalence of Coronavirus Disease 2019 in Egypt: Results of a community-based cohort. PLoS Pathog. 2021 Mar 11;17(3):e1009413. doi: 10.1371/journal.ppat.1009413. eCollection 2021 Mar. PMID 33705496
- [Result] Schmidt F, Weisblum Y, Muecksch F, Hoffmann HH, Michailidis E, Lorenzi JCC, Mendoza P, Rutkowska M, Bednarski E, Gaebler C, Agudelo M, Cho A, Wang Z, Gazumyan A, Cipolla M, Caskey M, Robbiani DF, Nussenzweig MC, Rice CM, Hatziioannou T, Bieniasz PD. Measuring SARS-CoV-2 neutralizing antibody activity using pseudotyped and chimeric viruses. J Exp Med. 2020 Nov 2;217(11):e20201181. doi: 10.1084/jem.20201181. PMID 32692348